CLINICAL TRIAL: NCT06291402
Title: Nasal Packing Duration and Its Role in the Development of Pharyngitis After Septorhinoplasty Surgery: A Prospective Observational Study
Brief Title: Nasal Packing Duration and Development of Pharyngitis After Septorhinoplasty Surgery
Status: Recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Other Study IDs: RC 34-1-2024
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Septoplasty or septal reconstruction is a corrective surgical procedure performed to straighten the nasal septum. It may be associated with numerous complications. To minimize these complications, both nasal cavities are frequently packed with different types of nasal packing. In our study we will try to find relationship between duration of nasal packing and postrhinoplasty sore throat and pharyngitis.

DETAILED DESCRIPTION:
Nasal packing affects swallowing by different mechanisms. It may affect swallowing as a result of nasal congestion, constant mouth breathing, throat dryness and pharyngitis.

Postoperative sore throat causes patient dissatisfaction and poor pain control. Several interventions could be performed to reduce sore throat and pharyngitis and increase patient satisfaction , which may not be convenient for all patients, such as gargling or sprays

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients
* aged from 20 to 40 years old
* undergo septorhinoplasty

Exclusion Criteria:

* Bleeding disorders
* Uncontrolled hypertension
* Cardiovascular diseases
* Uncontrolled diabetes mellitus
* Collagen disorders
* Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 ASA I and II patients aged from 20 to 40 years old will undergo septorhinoplasty in Benha university hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Sore throat | 48 hours postoperatively
  The incidence of Sore throat will be graded as 0 = Nil, 1 = Mild, 2 = Moderate and 3 = Severe as possible.

SECONDARY OUTCOMES:
Dysphagia | 48 hours postoperatively
  The incidence of Dysphagia will be recorded
Throat irritation | 48 hours postoperatively
  The incidence of throat irritation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Kohaf, ph.d, Principal Investigator — Al-Azhar University
Locations (1):
- Neveen Kohaf, Tanta, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request from the principle investigator
Supporting Information: Study Protocol, SAP